CLINICAL TRIAL: NCT03237494
Title: Genetic Screening of an At-risk Population for Hereditary TransthyRetin-related AMyloidosis and Longitudinal Monitoring of TTR Positive Subjects- A Multicenter Epidemiological Longitudinal Protocol
Brief Title: TRAMmoniTTR Study Genetic Screening of an At-risk Population for hATTR and Monitoring of TTR Positive Subjects
Acronym: TRAMmoniTTR
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: TRAM2 analysis
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-09

CONDITIONS: Transthyretin Amyloidosis; Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy; Transthyretin-Related (ATTR) Familial Amyloid Cardiomyopathy; Polyneuropathies; Cardiomyopathies
Keywords: Peripheral Nervous System Diseases; Transthyretin Amyloidosis; Transthyretin-related familial amyloid polyneuropathy; Transthyretin-related familial amyloid cardiomyopathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloid Neuropathies, Familial; Polyneuropathies; Cardiomyopathies; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants at risk for hATTR and participants diagnosed with hATTR: Participants 18 years of age or older

SUMMARY:
National, multicenter, epidemiological, longitudinal protocol to investigate the hATTR prevalence in an at-risk population for Hereditary Transthyretin Amyloidosis (hATTR) and subjects diagnosed with hATTR, to monitor the clinical status in TTR positive subjects and to establish hATTR biomarker/s

DETAILED DESCRIPTION:
Hereditary TransThyRetin Amyloidosis (hATTR) is a slowly progressive condition, that is transmitted as an autosomal dominant trait and is characterized by abnormal extracellular deposits of fibrillar, misfolded proteins (amyloid fibrils) in the body. Amyloid fibrils can be deposited in different body compartments, such as the nerves, heart, gastrointestinal tract, kidneys and brain, causing severe structural changes. More than 30 proteins can trigger the formation of amyloid fibrils, 5 of which can infiltrate the heart and cause cardiac amyloidosis.

One of these amyloidogenic protein is transthyretin, formerly known as prealbumin. Transthyretin (TTR) is found primarily in the serum (secreted by the liver) and cerebrospinal fluid (secreted by the choroid plexus) and functions as a carrier for the hormone thyroxine (T4) and retinol-binding protein (bound to retinol or vitamin A). The destabilization of the TTR protein and the formation of misfolded TTR.

It is the goal of this study to investigate the prevalence of Hereditary Transthyretin-related Amyloidosis (hATTR) in a cohort of 5.000 subjects are at risk for Hereditary Transthyretin Amyloidosis (hATTR) and subjects diagnosed with hATTR, to monitor the clinical status in TTR positive subjects and to establish hATTR biomarker/s.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant
* The participant is 18 years of age or older
* The participant has no diagnosis of alcoholism according to international guidelines
* The participant has not undergone chemotherapy for any carcinoma

AND

The participant is at risk for hATTR due to two or more the factors listed below:

* cardiomyopathy or polyneuropathy with no obvious etiology atypical Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) or Motor Neuron Disease (MND)
* autonomic dysfunction
* hypertrophic cardiomyopathy or heart failure with preserved ejection fraction Left Ventricular Hypertrophy (LVH)
* bilateral carpal tunnel syndrome
* spinal stenosis or spinal radiculopathy
* gait disorders
* ocular changes involving vitreous opacities
* unexplained weight loss >5kg
* renal abnormalities
* family history of hATTR
* based on imaging or biopsy suspected for the wild type TTR (ATTR) and not genetically tested for hATTR

OR • The participant is diagnosed with hATTR

OR

• The participant is a 1st or 2nd degree relative of the TTR positive subject

Exclusion Criteria

* Informed consent is not obtained from the participant
* The participant is younger than 18 years of age
* The participant has a diagnosis of alcoholism according to International guidelines
* The participant has undergone chemotherapy for any carcinoma
* The participant is not at risk for hATTR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at risk for Hereditary Transthyretin Amyloidosis (hATTR) and participants diagnosed with hATTR
Sampling Method: Probability Sample
Enrollment: 5028 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Analysis of prevalance of hATTR mutations among a cohort of participants at risk for hATTR. | 4 years
  DBS-based genetic analyses of TTR gene will be perfomed via the combination of the Next-Generation Sequencing (the mutation will be confirmed by Sanger sequencing) and the Multiplex ligation-dependent probe amplification.
To monitor clinical status in TTR positive subjects. | 4 years
  8 Follow up visits within 24 months

SECONDARY OUTCOMES:
Establishment of biomarker/s in TTR positive cohort. | 4 years
  hATTR-positive samples will be analyzed for the identification of potential biomarkers (based on MS/MS-Tandem spectroscopy) and compared with the merged control samples in order establish a HAE specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (84):
- Austria (2):
  - Kepler Universitätsklinikum, Klinik für Interne 1 - Kardiologie und internistische Intensivmedizin; Cardiology, Linz
  - Kepler Universitätsklinikum, Neuromed Campus; Neurology, Linz
- Germany (79):
  - Universitätsklinikum Aachen, Neurology, Aachen
  - Klinikum Westmünsterland GmbH, I. Medizinische Klinik und Interventionelle Kardiologie, Ahaus
  - Kreiskrankenhaus Altenburg, Neurology, Altenburg
  - Sächsisches Krankenhaus Arnsdorf, Akademisches Lehrkrankenhaus der TU Dresden, Neurology, Arnsdorf
  - Gemeinschaftspraxis Neurologie & Psychiatrie im Stadtpalais, Aschaffenburg
  - Kerckhoff-Klinik GmbH, Klinik für Kardiologie, Cardiology, Bad Nauheim
  - RHÖN-KLINIKUM Campus Bad Neustadt, Neurology, Bad Neustadt an der Saale
  - Charité - Universitätsmedizin Berlin Funktionsdiagnostik und Stationen, Cardiology, Berlin
  - Charité Universitätsmedizin Berlin, Klinik für Neurologie, Neurology, Berlin
  - Sana Klinikum Lichtenberg, Berlin
  - Charité Universitätsmedizin Berlin - Campus Virchow Klinikum (CVK), Cardiology, Berlin
  - Klinikum Bielefeld, Klinik für Kardiologie und internistische Intensivmedizin, Cardiology, Bielefeld
  - Evangelisches Klinikum Bethel gGmbH v. Bodelschwinghsche Stiftungen Bethel, Neurology, Bielefeld
  - Klinikum Bremen Mitte gGmbH, Neurologische Klinik, Neurology, Bremen
  - Gesundheit Nord gGmbH - Klinikverband Bremen, Bremen
  - Krankenhaus Buchholz und Winsen, gemeinnützige GmbH, Cardiology, Buchholz in der Nordheide
  - Krankenhaus Buchholz und Winsen, gemeinnützige GmbH, Neurology, Buchholz in der Nordheide
  - Allgemeines Krankenhaus Celle, Neurology, Celle
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - St. Vincenz Krankenhaus Datteln, Medizinische Klinik II, Cardiology, Datteln
  - Klinikum Dortmund gGmbH,Stroke-Unit und Neurologische Intensivstation, Neurology, Dortmund
  - LVR Klinikum Düsseldorf, Neurology, Düsseldorf
  - Martin Gropius Krankenhaus, Klinik für Neurologie, Neurology, Eberswalde
  - Universitätsklinikum Erlangen, Cardiology, Erlangen
  - Alfried Krupp Krankenhaus Rüttenscheid, Neurology, Essen
  - Contilia Herz- und Gefäßzentrum, Elisabeth-Krankenhaus Essen, Cardiology, Essen
  - Kliniken an der Paar Friedberg Krankenhaus, Cardiology, Friedberg
  - Herz-Thorax-Zentrum Fulda, Klinikum Fulda gAG, Universitätsmedizin Marburg - Campus Fulda, Cardiology, Fulda
  - University of Giessen-Marburg, Neurology, Giessen
  - Universitätsmedizin Göttingen - Herzzentrum; Cardiology, Göttingen
  - Universitätsklinikum Greifswald der Ernst-Moritz-Arndt-Universität, Neurology, Greifswald
  - kbo-Isar-Amper-Klinikum München-Ost, Klinik für Neurologie, Neurology, Haar
  - Martin-Luther-Universität, Universitätsklinik und Poliklinik für Neurologie, Neurology, Halle
  - Universitätsklinik und Poliklinik für Innere Medizin III, Cardiology, Halle
  - Asklepios Klinik St. Georg, Klinik für Neurologie, Hamburg
  - Universitäres Herzzentrum Hamburg, Klinik für Allgemeine und Interventionelle Kardiologie, Universitätsklinikum Hamburg-Eppendorf, Cardiology, Hamburg
  - Neurologie Neuer Wall, Fachärzte für Neurologie & Psychiatrie, Neurology, Hamburg
  - Albertinen-Krankenhaus, Cardiology, Hamburg
  - Asklepios Klinik Altona, Neurologische Abteilung mit überregionaler Stroke Unit, Neurophysiologie und Neurologischer Intensivmedizin, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Neurologie; Neurology, Hanover
  - Universitätsklinikum Heidelberg, Klinik für Kardiologie, Angiologie und Pneumologie, Cardiology, Heidelberg
  - Lausitzer Seenland Klinikum GmbH, Klinik für Neurologie, Neurology, Hoyerswerda
  - Universitätsklinikum Jena, Neurology, Jena
  - Universitätsklinikum Jena Klinik für Innere Medizin I, Jena
  - DRK-Kliniken Nordhessen gGmbH , Klinik für Neurologie und Klinische Neurophysiologie, Neurology, Kassel
  - Alexianer Krefeld GmbH, Krankenhaus Maria Hilf, Neurology, Krefeld
  - Universitaetsklinikum Leipzig, Neurology, Leipzig
  - Klinikum St. Georg gGmbH, Leipzig
  - Asklepios Fachklinikum Lübben, Neurology, Lubin
  - Universitäres Herzzentrum Lübeck, Medizinische Klinik II, Lübeck
  - Sana Kliniken Lübeck GmbH, Medizinische Klinik II, Lübeck
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - DRK Schmerz-Zentrum, Neurology, Mainz
  - Johannes Gutenberg-Universität Mainz, Klinik und Poliklinik für Neurologie; Neurology, Mainz
  - Diakonissen Speyer-Mannheim, Diakonissenkrankenhaus Mannheim, Neurology, Mannheim
  - Neckar-Odenwald Kliniken gGmbH, Kreiskrankenhaus Mosbach, Kardiologie der Klinik für Innere Medizin, Mosbach
  - Ökumenisches Hainich Klinikum gGmbH, Neurology, Mühlhausen
  - Friedrich-Baur-Institut, Neurologische Klinik und Poliklinik, Neurology, München
  - Kardiologie München Nord, Cardiology, München
  - Ludwig-Maximilians-Universität München, Klinikum Großhadern, Neurologische Klinik und Poliklinik & Deutsches Schwindel- und Gleichgewichtszentrum DSGZ, Neurology, München
  - Klinik und Poliklinik für Neurologie, Klinikum rechts der Isar, Technische Universität München, München
  - Praxis für Neurologie, Neurology, München
  - Ruppiner Kliniken GmbH,Hochschulklinikum der MHB, Neurology, Neuruppin
  - UKRB Universitätsklinikum Ruppin Brandenburg, Neuruppin
  - Kreiskrankenhaus Prignitz gGmbH, Neurology, Perleberg
  - Krankenhaus Barmherzige Brüder Regensburg, Klinik für Neurologie, Neurology, Regensburg
  - Universitätsklinikum Regensburg, Cardiology, Regensburg
  - Nordwest-Krankenhaus Sanderbusch gGmbH, Neurologische Klinik, Neurology, Sande
  - Sächsisches Krankenhaus Altscherbitz, Neurology, Schkeuditz
  - Jung-Stilling Klinikum Siegen, Diakonie Westfalen Süd Neuro, Neurogeriatrie, Neurology, Siegen
  - Elbe Klinikum Stade, Stade
  - Asklepios Fachklinikum Teupitz, Neurology, Teupitz
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - NeuroPoint, Neurology, Ulm
  - University of Ulm, Neurology, Ulm
  - Sophien-u.Hufeland-Klinikum, Klinik für Neurologie und Klinische Neurophysiologie, Neurology, Weimar
  - Fachkrankenhaus Hubertusburg gGmbH, Neurologische Klinik, Neurology, Wermsdorf
  - Sana HANSE Klinikum Wismar, Klinik für Neurologie, Neurology, Wismar
  - Praxis für Neurologie, Neurology, Wolfratshausen
- Switzerland (3):
  - Luzerner Kantonspital, Cardiology, Lucerne
  - Solothurner Spitäler AG, Bürgerspital Solothurn, Cardiology, Olten
  - Praxisgemeinschaft für Kardiologie, Innere Medizin und Psychosomatische Medizin, Cardiology, Zug